CLINICAL TRIAL: NCT01722357
Title: Promoting Physical Activity Among Bariatric Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascension St. Vincent Carmel Hospital (Other)
Collaborators: St. Vincent Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09110
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Obesity
Keywords: bariatric surgery; physical activity; morbid obesity
MeSH Terms: conditions — Obesity; Motor Activity; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pedometer + Exercise Counseling (Experimental)
  Interventions: Behavioral: Pedometer; Behavioral: Exercise Counseling
- Pedometer (Experimental)
  Interventions: Behavioral: Pedometer
- Usual Care (No Intervention): Self-help information provided on physical activity (WIN:Weight Control Network "Active At Any Size" provided by National Institute of Diabetes and Digestive and Kidney Diseases, 2006).

INTERVENTIONS:
Behavioral: Pedometer — Participants are provided with Omron Model HJ-151 pedometers and given instruction on how to use the pedometer to set goals for increasing physical activity. They are given diaries to track their daily step counts.
  Arms: Pedometer; Pedometer + Exercise Counseling
Behavioral: Exercise Counseling — Manualized cognitive behavioral treatment program including goal setting, adding exercise throughout the day, physical limitations/injuries, maintaining motivation, benefits of exercise, FITT principles, exercise as recreation, and restructuring thoughts related to activity.
  Arms: Pedometer + Exercise Counseling

SUMMARY:
The purpose of the study is to address 3 main sets of questions in the bariatric surgery population. 1) Does bariatric surgery, without any other intervention, lead to increased physical activity and improved physical fitness? 2) Does wearing a pedometer lead to increased physical activity in obese individuals prior to and/or after bariatric surgery? Does the increased activity result in improvements in physical fitness? 3) Does physical activity counseling increase physical activity prior to and or/after bariatric surgery? Does the increased activity result in improvements in physical fitness? The overall goal of the study is to determine the impact of bariatric surgery on physical activity and assess the utility of additional interventions to help postoperative patients adopt a more active lifestyle. Participants are randomized to usual care, pedometer use, or pedometer use plus exercise counseling before and for the first 6 months after bariatric surgery. In an extension of the primary study, from 1 to 5 years after surgery, all patients receive exercise counseling. Physiological measures will be assessed to determine whether bariatric surgery and/or improved physical activity levels result in improved physical fitness.

DETAILED DESCRIPTION:
Bariatric surgery leads to improvement or resolution of a variety of health conditions. It is also well established that physical activity, with or without weight loss, improves many health-related problems and can have a positive impact on mood. Therefore, physical activity may amplify the health and psychological benefits often experienced from bariatric surgery. Prior to surgery many patients are relatively inactive due to physical and social barriers associated with their weight. In addition, many patients find it difficult to adopt an active lifestyle after surgery, despite an increased capacity to exercise. However, weight loss is associated with physical activity after bariatric surgery. Nonetheless, little is known about the most effective means to promote activity among this group of individuals. This study will examine changes in physical activity and fitness after bariatric surgery and examine whether the addition of pedometer use and exercise counseling may lead to greater improvements.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients planning to undergo bariatric surgery at the St. Vincent Bariatric Center of Excellence
* Men and women 18 years and older
* The participant must be motivated to enroll in a study assessing physical activity before and after bariatric surgery, able to understand and comply with the study, and must agree to return for scheduled visits
* All participants must sign a written, informed consent

Exclusion Criteria:

* History of myocardial infarction within the past three months, unstable angina pectoris, sustained or episodic cardiac arrhythmias that could be aggravated by physical activity, symptomatic peripheral vascular disease, or any other medical condition that the medically responsible investigator deems inappropriate.
* Abnormal electrocardiogram (ECG), assessed at the pretreatment screening visit that the medically responsible investigator deems inappropriate for participation in a physical activity program.
* Unable to progress toward 30 minutes of continuous walking during the 6 months of study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Accelerometer-Derived Activity | 6 months post-surgery
  accelerometer-derived activity will be collected.

SECONDARY OUTCOMES:
Graded Treadmill Test | baseline, 6 months and 5 years post-surgery
  length of time participant walks on treadmill until reaching percieved exertion or heart rate target
Upper Body Strength testing | baseline, 6 months and 5 years post-surgery
  hand grip and chest press
Baecke Habitual Physical Activity Questionnaire | baseline, 2, 4, 6, 12, and 18 months and 2, 3, 4, and 5 years post-surgery
Myers-Roth Benefits and Barriers of Exercise Questionnaire | baseline, 2, 4, 6, 12, and 18 months and 2, 3, 4, and 5 years post-surgery
PHQ-9 Symptom Checklist | baseline, 2, 4, 6, 12, and 18 months and 2, 3, 4, and 5 years post-surgery
  measure of depressed mood
St.Vincent Exercise Questionnaire | baseline , 2, 4, 6, 12, and 18 months and 2, 3, 4, and 5 years post-surgery
Exercise Identity Scale | 12 and 18 months, and 2, 3, 4, and 5 years post-surgery
NEO-IPIP Conscientiousness Scale | 12 and 18 months, and 2, 3, 4, and 5 years post-surgery
Thoughts of Exercise Scale | 12 and 18 months, and 2, 3, 4, and 5 years post-surgery
Accelerometer-Derived Activity | baseline, 2, 4, 6, 12, and 18 months and 2, 3, 4, and 5 years post-surgery

OTHER OUTCOMES:
Vital signs | baseline, 2, 4, 6, 12, and 18 months and 2, 3, 4, and 5 years post-surgery
  weight, blood pressure, pulse, respiratory rate

CONTACTS AND LOCATIONS:
Overall Officials: David B Creel, PhD, Principal Investigator — St. Vincent Carmel Hospital Bariatric Center of Excellence
Locations (1):
- St. Vincent Carmel Hospital Bariatric Center of Excellence, Carmel, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Creel DB, Schuh LM, Reed CA, Gomez AR, Hurst LA, Stote J, Cacucci BM. A randomized trial comparing two interventions to increase physical activity among patients undergoing bariatric surgery. Obesity (Silver Spring). 2016 Aug;24(8):1660-8. doi: 10.1002/oby.21548. Epub 2016 Jul 1. PMID 27367821
- [Derived] Creel DB, Schuh LM, Newton RL Jr, Stote JJ, Cacucci BM. Exercise Testing Reveals Everyday Physical Challenges of Bariatric Surgery Candidates. J Phys Act Health. 2017 Dec 1;14(12):913-918. doi: 10.1123/jpah.2017-0128. Epub 2017 Oct 12. PMID 28682736